CLINICAL TRIAL: NCT07129525
Title: Health Oriented Protocol for Epidermal Radiodermatitis,A Prospective Observational Study
Brief Title: Health Oriented Protocol for Epidermal Radiodermatitis
Acronym: HOPE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7545
Record Dates: First submitted 2025-07-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Pelvic Cancer; Radiation Skin Injury; Gynecologic Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Head and Neck Neoplasms; Pelvic Neoplasms; Radiation Injuries | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiation therapy — Patients treated with radiotherapy will be evaluated within a period of five to seven weeks, during which time radiation-induced skin toxicities will be assessed.

SUMMARY:
Radiation therapy is a standard treatment for malignant tumors of the head and neck and pelvic regions, used alone or in combination with chemotherapy. While effective, it is often associated with adverse effects that can impact patient outcomes. Among the most frequent toxicities is radiation-induced dermatitis (RID), affecting up to 95% of patients. These skin reactions, ranging in severity, may compromise quality of life and lead to treatment interruptions.The severity of RID is influenced by both intrinsic and extrinsic factors. Intrinsic factors include age, sex, ethnicity, nutritional status, and comorbidities such as diabetes or systemic inflammation. Extrinsic factors include the radiation technique, total dose, treated volume, and presence of infections. These variables require close monitoring to reduce complications.Radiation damages the skin and underlying tissues, causing xerosis, pigmentation changes, loss of elasticity, fibrosis, and varying degrees of dermatitis. Effective prevention starts with patient education and skincare support throughout treatment to reduce incidence and severity.In Italy, head and neck cancers, though less common than other malignancies, present a significant clinical burden. Laryngeal cancer accounts for around 5,000 new cases annually. Oral cavity, pharyngeal, and thyroid tumors also have notable incidence and require complex treatments such as (chemo)radiotherapy, increasing the risk of RID.RID represents not only a clinical issue but also a psychological and functional challenge. Pain, emotional distress, and reduced autonomy are key aspects affecting patients' overall wellbeing. A multidimensional approach that integrates clinical care and psychosocial support is essential.This study aims to investigate the relationship between RID severity, pain, psychological distress, and functional autonomy during radiotherapy or chemoradiotherapy, identifying predictors of severe toxicity and guiding personalized supportive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* with head and neck or pelvic malignancies
* undergoing either exclusive radiotherapy or concurrent chemoradiotherapy will be included, following signed informed consent.

Exclusion Criteria:

* Pediatric patients,
* patients with malignancies outside the head and neck or pelvic regions,
* patients who have not yet started or have already completed exclusive radiotherapy or concurrent chemoradiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with head and neck or pelvic malignancies undergoing either exclusive radiotherapy or concurrent chemoradiotherapy will be included
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of radiation-induced dermatitis | 5-7 weeks from treatment initiation
  Proportion of patients undergoing radiotherapy or chemoradiotherapy for head and neck or pelvic cancers who develop radiation-induced dermatitis, assessed according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
  Unit of Measure: % of patients with grade ≥1 dermatitis
Severity of radiation-induced dermatitis | 5-7 weeks from treatment initiation
  Maximum grade of radiation-induced dermatitis in patients undergoing radiotherapy or chemoradiotherapy for head and neck or pelvic cancers, assessed according to the CTCAE v5.0.
  Unit of Measure: CTCAE grade (0-5)

SECONDARY OUTCOMES:
Temporal evolution of dermatitis severity | 5-7 weeks from treatment initiation
  Change in toxicity grade of radiation-induced dermatitis across weekly assessments during radiotherapy or chemoradiotherapy, measured according to the CTCAE v5.0.
  Unit of Measure: Change in CTCAE grade (0-5) over time
Correlation between dermatitis severity and pain | 5-7 weeks from treatment initiation
  Correlation between dermatitis severity (CTCAE v5.0) and pain intensity (assessed with the Numeric Rating Scale, 0-10).
  Unit of Measure: Correlation coefficient (r)
Correlation between dermatitis severity and psychological distress | 5-7 weeks from treatment initiation
  Correlation between dermatitis severity (CTCAE v5.0) and psychological distress (assessed with the Distress Thermometer - DT).
  Unit of Measure: Correlation coefficient (r)
Correlation between dermatitis severity and functional autonomy | 5-7 weeks from treatment initiation
  Correlation between dermatitis severity (CTCAE v5.0) and functional autonomy (assessed with the Barthel Index).
  Unit of Measure: Correlation coefficient (r)

CONTACTS AND LOCATIONS:
Overall Officials: danilo pasini, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS